CLINICAL TRIAL: NCT05980494
Title: Validity of Lung Ultrasound Score and Inferior Vena Cava Diameter Compared to Pulse Pressure Variation Predicting Fluid Responsiveness in Mechanically Ventilated Critically Ill Patients: a Comparative Study
Brief Title: Lung Ultrasound Score and Inferior Vena Cava Diameter Compared to Pulse Pressure Variation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Hamed, Associate professor, Fayoum University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: D 310
Record Dates: First submitted 2023-07-31; First posted 2023-08-08 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Sepsis; Critical Illness
Keywords: lung utlrasound; pulse pressure variation; inferior vena cava; fluid responsiveness
MeSH Terms: conditions — Sepsis; Critical Illness | interventions — Saline Solution

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Scanning group (Experimental): Lung ultrasound (LUS), Inferior vena cava ultrasound (IVC US) and pulse pressure variation (PPV) will be done to every patient in the study.
  Interventions: Drug: normal Saline; Device: lung ultrasound; Device: inferior vena cava measurements; Diagnostic Test: passive leg raising test (PLRT); Device: pulse pressure variation

INTERVENTIONS:
Drug: normal Saline — normal saline cyrstalloids infusion with rate of 4ml/kg /h for 3 hours
  Other Names: Fluid challenge test
Device: lung ultrasound — Lung ultrasound by Philips clear vue350, Philips healthcare, Andover MAO1810, USA, Machine ID:1385 will scan For each hemi-thorax 3 main areas (anterior (Ant), lateral (Lt) and posterior (Post)) marked by the para-sternal, anterior axillary and posterior axillary lines for a total of 28 sectors will be identified
Device: inferior vena cava measurements — The inferior vena cava was explored in the subxiphoid window in its sagittal view-just below the junction between the inferior vena cava and suprahepatic veins which lie approximately 0.5 to 3 cm from the right atrium, following the American Society of Echocardiography guidelines.; The (IVC distensibility index (dIVC) was calculated as (maximum diameter - minimum diameter)/minimum diameter.
Diagnostic Test: passive leg raising test (PLRT) — Regardless of CVP (i.e., during "blind PLR"), noninvasiveΔPLR systolic arterial pressure (SAP) more than 17% reliably identify fluid responders. During "CVP-guided PLR", in case of sufficient change in CVP (at least of 2 mmHg), noninvasiveΔPLR SAP perform better (cutoff of 9%). These findings, in sedated patients who had already undergone volume expansion and/or catecholamines, have to be verified during the early phase of circulatory failure (before an arterial line).
Device: pulse pressure variation — patients will be temporarily sedated and paralyzed and on fully controlled mechanical ventilation. No spontaneous breathing effort will be detected on the mechanical ventilator waveform monitor ensuring that the respiratory changes in arterial pressure reflected only the effects of positive pressure ventilation. Modes of ventilation is selected to volume or pressure controlled ventilation, depending on the decision of the primary physicians. A tidal volume will be not less than 8 ml/ kg (predicted body weight). The preset respiratory rate will be at 14 breath/min. Positive end expiratory pressure (PEEP) will be between 8 and 10 cmH2O. The plateau pressure was kept at below 30 cmH2O. In all patients, radial artery cannulation will be done for invasive blood pressure monitoring (using a 20 G cannula), PPV is calculated directly on Nihon Kohden monitores at base line.

SUMMARY:
Evaluation and management of intravascular volume are a central challenge for the critical ill patients. Hypotensive patients are commonly resuscitated with intravenous crystalloid fluid as a recommendation for treatment of many shock states.

There has been a growing interest in the implementation of lung ultrasound in critical care management in the last decade as it is easy, bedside, non-expensive, non invasive and radiation free.

The object of the current study is to assess the ability of lung and inferior vena cava sonography versus pulse pressure variation to predict fluid responsiveness in patients with circulatory failure on mechanical ventilation.

DETAILED DESCRIPTION:
The study will be conducted in intensive care units of Fayoum University Hospitals after approval of the local institutional ethics committee and local institutional review board. Hypotensive Patients on mechanical ventilation starting from August 2022 will be enrolled in this prospective study until fulfilling sample size. A detailed informed consent will be signed before recruitment. All patients who fulfilled inclusion criteria will be monitored by: 6 leads ECG, Blood pressure, Urinary catheter for urine output, Pulse oximter.Lung ultrasound (LUS), Inferior vena cava ultrasound (IVC US) and pulse pressure variation (PPV) will be done to every patient in the study. The Consolidated standards of Reporting Trials (CONSORT) recommendation will be followed. LUS and IVC measurements were performed by using a convex ultrasound probe (Philips clear vue350, Philips healthcare, Andover MAO1810, USA, Machine ID: 1385). LUS will be performed by an experienced radiologist according to standardized protocols. For each hemi-thorax 3 main areas (anterior (Ant), lateral (Lt) and posterior (Post)) marked by the para-sternal, anterior axillary and posterior axillary lines for a total of 28 sectors will be identified. Each one will be divided into upper and lower halves, making a sum of 6 different quadrants for each side: anterior superior, anterior inferior, lateral superior, lateral inferior, posterior superior, posterior inferior. Ultrasound examination of the anterolateral chest was carried out with longitudinal scan of the right and left hemi thoraces, from the second to the fourth (on the right side to the ﬁfth) intercostal space, as previously described. For each quadrant a score will be assigned based on B lines which are defined as an echogenic artifact with a narrow origin on the pleural line, deepening to the inferior border of the screen and coherent with respiratory movements indicating subpleural interstitial edema as follows:

(0) Normal aeration: A lines with lung sliding or fewer than two isolated B lines

1. Moderate loss of lung aeration: well-defined, multiple B lines.
2. Severe loss of lung aeration: multiple coalescent B lines.
3. Complete loss of lung aeration or lung consolidation. This will be used to calculate total LUS-score (calculated as a sum of all quadrants score) and individual areas score (Ant, Lt and Post).

IVC US: The inferior vena cava was explored in the subxiphoid window in its sagittal view-just below the junction between the inferior vena cava and suprahepatic veins which lie approximately 0.5 to 3 cm from the right atrium, following the American Society of Echocardiography guidelines.; The (IVC distensibility index (dIVC) was calculated as (maximum diameter - minimum diameter)/minimum diameter.

PPV: patients will be temporarily sedated and paralyzed and on fully controlled mechanical ventilation. No spontaneous breathing effort will be detected on the mechanical ventilator waveform monitor ensuring that the respiratory changes in arterial pressure reflected only the effects of positive pressure ventilation. Modes of ventilation is selected to volume or pressure controlled ventilation, depending on the decision of the primary physicians. A tidal volume will be not less than 8 ml/ kg (predicted body weight). The preset respiratory rate will be at 14 breath/min. Positive end expiratory pressure (PEEP) will be between 8 and 10 cmH2O. The plateau pressure was kept at below 30 cmH2O. In all patients, radial artery cannulation will be done for invasive blood pressure monitoring (using a 20 G cannula), PPV is calculated directly on Nihon Kohden monitores at base line.

• Sample size: Sample size was calculated using MedCalc Statistical Software version 20 (MedCalc Software, Ostend, Belgium. Minimal sample size of patients was 118 patients with 59 responsive cases and 59 non-responsive cases. Calculation is guided by AUC of 0.915 obtained from a study in comparison to a null value of 0.8, with alpha of 0.05 and power of 90%. Sample size will be increased to 150 patients to increase precision and ensure that at least 59 responsive and 59 non-responsive cases are included.

• Statistical analysis: Data will be collected and coded using Microsoft Excel and data analysis will be performed using IBM SPSS version 28 for Windows. Descriptive statistics will be presented in the form of numbers and percentages of categorical data, while means with standard deviations or medians with interquartile ranges will be used for numerical data variables. ROC curve will be used to estimate the appropriate cut off point for the inferior vena cava distensibility index, and for the lung ultrasound score. Area under the curve (AUC) will be reported and will be used to compare the diagnostic ability of different tests. Sensitivity, specificity, positive predictive value and negative predictive value will be reported with the 95% confidence intervals. P-value < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients on mechanical ventilation (MV).
* Aged more than 18 years.
* Mean arterial pressure (MAP) less than 65 mmHg or systolic arterial pressure less than 90mm Hg with signs of hypoperfusion (urinary flow < 0.5mL/kg/ h for > 2hr , tachycardia > 100 beats/min, or presence of skin mottling , and seurm lactate more than 2 mmol/L).

Exclusion Criteria:

* Cardiac arrhythmias.
* Previously known significant valvular disease or intracardiac shunt.
* Chest drains.
* Increasing intra abdominal pressure.
* Prephiral vascular disesaes.
* Adult respiratory distress syndrome (ARDS) patients due to low tidal volume.
* Interstitial lung disease because B-lines in these conditions are the consequence of the thickened interlobular septa characterizing ﬁbrosis and are not modiﬁed by the state of hydration or imbibition 12
* Any contraindication for fluid administration as cardiogenic shock, acute pulmonary edema or LVEF% less than 50%.
* Renal patients with oliguria and volume overload including patients on hemodialysis or patients with acute anuric renal failure.
* Patients with lower extremity artery/vein thrombosis, significant lower extremity artery plaque, lower extremity artery occlusion, inferior vena cava filter implantation and lower extremity varicose veins.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
The sensitivity of lung ultrasound in predicting fluid responsiveness. | After 5 minutes of admission
  <0.8: non-sensitive, >0.8: sensitive

SECONDARY OUTCOMES:
lung ultrasound B lines score | after 5 minutes of admission
  (0) Normal aeration: A lines with lung sliding or fewer than two isolated B lines
  1. Moderate loss of lung aeration: well-defined, multiple B lines.
  2. Severe loss of lung aeration: multiple coalescent B lines.
  3. Complete loss of lung aeration or lung consolidation. This will be used to calculate total LUS-score (calculated as a sum of all quadrants score) and individual areas score (Ant, Lt and Post).
Inferior vena cava distensibility index. | after 10 minutes of admission
  (maximum diameter - minimum diameter)/minimum diameter.
pulse pressure variation | 15 minutes after admission
  in percent
central venous pressure | after 20 minutes of admission
  in centimeter water
heart rate | 5 minutes after admission
  in beat per minute
serum lactate | after 30 minutes of admission
  in ml equivalent per liter
urine output | in 1 hour after admission
  in ml/ hour
length of stay in ICU | 1 hour after discharge
  in days
specificity of lung ultrasound predicting fluid responsiveness | 5 minutes after admission
  <0.8 non specific > 0.8 specific
sensitivity of IVC ultrasound predicting fluid responsiveness | after 5 minutes of admission
  <0.8 non sensitive >0.8 sensitive
sensitivity of pulse pressure variation predicting fluid responsiveness | after 5 minutes of admission
  <0.8 non sensitive >0.8 sensitive
specificity of IVC ultrasound predicting fluid responsiveness | after 5 minutes of admission
  <0.8 non sensitive >0.8 sensitive
specificity of pulse pressure variation predicting fluid responsiveness | after 5 minutes of admission
  <0.8 non sensitive >0.8 sensitive

OTHER OUTCOMES:
weight | 5 minutes before admission
  in kilogram
height | 5 minutes before admission
  in centimeters
body mass index | 5 minutes before admission
  in kilogram/m2
age | 5 minutes before admission
  in years

CONTACTS AND LOCATIONS:
Overall Officials: omar S farghaly, MD, Study Director — lecturer
Locations (1):
- Fayoum University Hospital, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chvojka J, Matejovic M. [International guidelines for management of severe sepsis and septic shock 2012 - comment]. Vnitr Lek. 2014 Jan;60(1):59-67. Czech. PMID 24564777
- [Background] Haddam M, Zieleskiewicz L, Perbet S, Baldovini A, Guervilly C, Arbelot C, Noel A, Vigne C, Hammad E, Antonini F, Lehingue S, Peytel E, Lu Q, Bouhemad B, Golmard JL, Langeron O, Martin C, Muller L, Rouby JJ, Constantin JM, Papazian L, Leone M; CAR'Echo Collaborative Network; AzuRea Collaborative Network. Lung ultrasonography for assessment of oxygenation response to prone position ventilation in ARDS. Intensive Care Med. 2016 Oct;42(10):1546-1556. doi: 10.1007/s00134-016-4411-7. Epub 2016 Jun 20. PMID 27324241